CLINICAL TRIAL: NCT04596137
Title: Kangaroo Care Reduces Infant Pain Caused By Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, DENİZ YİĞİT, Research Assistant, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DYIGIT2; Emel SEZICI (Other: Kütahya Health Sciences University)
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Infant; Pain; Kangaroo Mother Care; Nursing; Evidence-based Practices
Keywords: infant; pain; kangaroo mother care; nursing; evidence-based practices
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted between May -September 2016 in FHC. As 1-month-old infants were enrolled for the study, the total number of infants enrolled in FHCs each month was determined. Post-natal infants numbers were recorded in May-June, June-July, July-August, and August-September, for 48, 52, 59, and 57 infants, respectively. A pilot study was conducted on 20 infants born in May. Following the pilot study, monthly randomization was performed by an investigator. Accordingly, the study and control groups were determined monthly. There was no blinding in this study.
Masking Description: Researchers and family of infants knew about all the details of the study. Verbal and written permission was obtained from families.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- İnfant pain management (Experimental): Kangaroo mother care was applied to the infants during heel prick. With kangaroo mother care, the pain of infants was reduced.
  Interventions: Behavioral: İnfant pain management

INTERVENTIONS:
Behavioral: İnfant pain management — Kangaroo mother care was applied to the infants during heel prick. With kangaroo mother care, the pain of infants was reduced.

SUMMARY:
The aim of this randomized controlled study determine the effect of KMC on pain in infants during vaccination.

DETAILED DESCRIPTION:
Infants undergo many painful procedures from the time they are born. Kangaroo mother care (KMC) is one of the nonpharmacological methods that are effective in alleviating pain. The aim of this randomized controlled study determine the effect of KMC on pain in infants during vaccination. The study subjects were 128 healthy, 1-month-old infants and their mothers. A sociodemographic questionnaire, the Neonatal Infant Pain Scale (NIPS), a pulse oximeter, and a chronometer were used in collecting the data. This study indicate that KMC reduced crying duration, heart rate, and pain in vaccinated infants, whereas it increased oxygen saturation levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* The consent of the parents to participate in the application of the study,
* The infant being 1 month old
* Parents and infants being healthy

Exclusion Criteria:

* The consent of the parents not to participate in the application of the study,
* The infant not being 1 month old
* The parents and infants not being healthy.

Ages: 1 Minute to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Pain control of infants | during 5 minutes
  The infant's pain was reduced by applying kangaroo mother care during the heel blood collection of infants.Pain level was determined with the pain scale. Pain score decreased at the end of the application.

SECONDARY OUTCOMES:
Reduce crying time of infants | during 5 minutes
  Crying time of infants decreased with kangaroo mother care applied during heel prick.
Control heart rate of infants | during 5 minutes
  With kangaroo mother care applied during the heel prick, the heart rate of the babies was kept under control.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz YİĞİT, Res.Asst., Principal Investigator — ESOGÜ

IPD SHARING:
Plan to Share IPD: Yes
Other researchers can access the entire article.
Supporting Information: Study Protocol
Time Frame: They can reach constantly
Access Criteria: Being a healthcare professional working with infants

REFERENCES:
- [Result] Buyukgonenc L, Toruner EK. Pain and nursing management in childhood. In: Conk Z, Başbakkal Z, Bal Yılmaz H, Bolışık B, eds. Pediatric Nursing (pp.881-889). Ankara: Academician Bookstore; 2013.
- [Result] Johnston C, Campbell-Yeo M, Fernandes A, Inglis D, Streiner D, Zee R. Skin-to-skin care for procedural pain in neonates. Cochrane Database Syst Rev. 2014 Jan 23;(1):CD008435. doi: 10.1002/14651858.CD008435.pub2. PMID 24459000
- [Result] Kostandy R, Anderson GC, Good M. Skin-to-skin contact diminishes pain from hepatitis B vaccine injection in healthy full-term neonates. Neonatal Netw. 2013 Jul-Aug;32(4):274-80. doi: 10.1891/0730-0832.32.4.274. PMID 23835546
- [Result] Witt N, Coynor S, Edwards C, Bradshaw H. A Guide to Pain Assessment and Management in the Neonate. Curr Emerg Hosp Med Rep. 2016;4:1-10. doi: 10.1007/s40138-016-0089-y. Epub 2016 Mar 12. PMID 27073748
- [Result] Choudhary M, Dogiyal H, Sharma D, Datt Gupta B, Madabhavi I, Choudhary JS, Choudhary SK. To study the effect of Kangaroo Mother Care on pain response in preterm neonates and to determine the behavioral and physiological responses to painful stimuli in preterm neonates: a study from western Rajasthan. J Matern Fetal Neonatal Med. 2016 Mar;29(5):826-31. doi: 10.3109/14767058.2015.1020419. Epub 2015 Mar 18. PMID 25758623
- [Result] Hartley KA, Miller CS, Gephart SM. Facilitated tucking to reduce pain in neonates: evidence for best practice. Adv Neonatal Care. 2015 Jun;15(3):201-8. doi: 10.1097/ANC.0000000000000193. PMID 26002861
- [Result] Asadi-Noghabi F, Tavassoli-Farahi M, Yousefi H, Sadeghi T. Neonate pain management: what do nurses really know? Glob J Health Sci. 2014 Jul 14;6(5):284-93. doi: 10.5539/gjhs.v6n5p284. PMID 25168978
- [Result] Conde-Agudelo A, Diaz-Rossello JL. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2016 Aug 23;2016(8):CD002771. doi: 10.1002/14651858.CD002771.pub4. PMID 27552521
- [Result] Moore ER, Bergman N, Anderson GC, Medley N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2016 Nov 25;11(11):CD003519. doi: 10.1002/14651858.CD003519.pub4. PMID 27885658
- [Result] Cho ES, Kim SJ, Kwon MS, Cho H, Kim EH, Jun EM, Lee S. The Effects of Kangaroo Care in the Neonatal Intensive Care Unit on the Physiological Functions of Preterm Infants, Maternal-Infant Attachment, and Maternal Stress. J Pediatr Nurs. 2016 Jul-Aug;31(4):430-8. doi: 10.1016/j.pedn.2016.02.007. Epub 2016 Mar 11. PMID 26975461
- [Result] Kostandy RR, Ludington-Hoe SM. Clustered pain procedures in skin-to-skin contact (ssc) position for full term newborns. World. 2017;7:38-47. Doi: 10.4236/wjns.2017.71004.
- [Result] Bera A, Ghosh J, Singh AK, Hazra A, Som T, Munian D. Effect of kangaroo mother care on vital physiological parameters of the low birth weight newborn. Indian J Community Med. 2014 Oct;39(4):245-9. doi: 10.4103/0970-0218.143030. PMID 25364150
- [Result] Sutar R, Baraha S, Mummidi PS. Effects of kangaroo mother care on common vital parameters of preterm infants. Int J Sci Res. 2015;4(12):373-375.
- [Result] World Health Organization (WHO) (2003). Kangaroo mother care: A practical guide. Available at https://www.who.int/maternal_child_adolescent/documents/9241590351/en/. Accessed February 18, 2019.
- [Result] Saeidi R, Asnaashari Z, Amirnejad M, Esmaeili H, Robatsangi MG. Use of "kangaroo care" to alleviate the intensity of vaccination pain in newborns. Iran J Pediatr. 2011 Mar;21(1):99-102. PMID 23056772
- [Result] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Result] Akdovan T, Yıldırım, Z. Assessment of pain in healthy neonates, investigation of the effects of pacifying and holding in the arms [master dissertation]. Istanbul: Health Sciences Institute; 1999.
- [Result] Akyurek B, Conk Z. 2006. Examining the effectiveness of nonpharmacological pain-reducing methods in newborns during needle-based procedures. J Ege Univ Sch Nurs. 2006;22(1):1-17.
- [Result] Okan F, Ozdil A, Bulbul A, Yapici Z, Nuhoglu A. Analgesic effects of skin-to-skin contact and breastfeeding in procedural pain in healthy term neonates. Ann Trop Paediatr. 2010;30(2):119-28. doi: 10.1179/146532810X12703902516121. PMID 20522298
- [Result] Gray L, Watt L, Blass EM. Skin-to-skin contact is analgesic in healthy newborns. Pediatrics. 2000 Jan;105(1):e14. doi: 10.1542/peds.105.1.e14. PMID 10617751
- [Result] Nimbalkar SM, Chaudhary NS, Gadhavi KV, Phatak A. Kangaroo Mother Care in reducing pain in preterm neonates on heel prick. Indian J Pediatr. 2013 Jan;80(1):6-10. doi: 10.1007/s12098-012-0760-6. Epub 2012 Apr 28. PMID 22544676
- [Result] Kashaninia Z, Sajedi F, Rahgozar M, Noghabi FA. The effect of Kangaroo Care on behavioral responses to pain of an intramuscular injection in neonates. J Spec Pediatr Nurs. 2008 Oct;13(4):275-80. doi: 10.1111/j.1744-6155.2008.00165.x. PMID 19238715
- [Result] Dezhdar S, Jahanpour F, Firouz Bakht S, Ostovar A. The Effects of Kangaroo Mother Care and Swaddling on Venipuncture Pain in Premature Neonates: A Randomized Clinical Trial. Iran Red Crescent Med J. 2016 Feb 21;18(4):e29649. doi: 10.5812/ircmj.29649. eCollection 2016 Apr. PMID 27274399
- [Result] Stuard W. The effects of kangaroo care on a newborn development and vital physiology. Clin Mother Child Health. 2016;13(1):1-4. Doi: 10.4172/2090-7214.1000225.
- [Result] Moore ER, Anderson GC, Bergman N, Dowswell T. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2012 May 16;5(5):CD003519. doi: 10.1002/14651858.CD003519.pub3. PMID 22592691